CLINICAL TRIAL: NCT05834556
Title: Home-based Prehabilitation for Frail Cardiac Surgery Patients (HOME FREE) - A Quasi-experimental Feasibility Study
Brief Title: Home-based Exercise for Frail Individuals Prior to Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Todd A Duhamel (Other)
Responsible Party: Sponsor-Investigator, Dr. Todd A Duhamel, Professor, Faculty of Kinesiology and Recreation Management, St. Boniface Hospital
Organization: St. Boniface Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOME FREE
Record Dates: First submitted 2023-03-24; First posted 2023-04-28 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Frailty; Pre-operative Exercise; Prehabilitation; Cardiac Surgery; Telerehabilitation
Keywords: telerehabilitation; prehabilitation; cardiac surgery; frailty; pre-operative exercise
MeSH Terms: conditions — Frailty | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation group (Experimental): Participants will engage in 4 virtual sessions with a physiotherapist, over a 3 week period. They will be prescribed an individual exercise program (based on assessment). Participants will complete the program 3x/week independently and diarize the exercise on provided documents. For participants living within Winnipeg, they will also diarize their accelerometer use/sleeping times during wear.
  Interventions: Behavioral: Prehabilitation

INTERVENTIONS:
Behavioral: Prehabilitation — Everyone will participate in a home-based prehab program with individual video sessions with a physiotherapist at 4 time points over a period of 3 weeks. The initial session will take an hour and consist of a subjective and physical assessment followed by an individualized exercise program demonstration and education. Patients will be instructed to complete the exercises independently 3x/week. The second and third sessions will be 30 minutes in duration and will check in on activity progress, the presence of abnormal responses to exercise, review exercise technique, address barriers and facilitators to activity completion as well as provide support and encouragement for the current level of activity. The final session will take 30 minutes and will review exercise progress, presence of abnormal responses to exercise followed by a reassessment of physical function.

SUMMARY:
The goal of this quasi-experimental feasibility study is to determine if a home based exercise program, that is supported virtually by a physiotherapist, is feasible for frail adults that are waiting for cardiac surgery. The main questions it aims to answer are:

* Will patients be interested in participating in a virtual home-based exercise program before surgery?
* Is the prescribed program practical? Will participants complete the exercises as prescribed, 3x/week?
* Are the exercise images, videos, and live, virtual sessions with the physiotherapists good enough to allow the participant to be independent with good exercise technique?
* Are the 4 virtual sessions able to be done in the specified time frames (1hr initial assessment, 30 minute follow ups)?
* Can the exercise program be done with out any major adverse events?
* What are the physical activity behaviours of frail participants awaiting cardiac surgery? Do they improve with an exercise program?

Participants will be required to:

* meet with a physiotherapist virtually (Zoom or Microsoft Teams) 4 times over a 3 week period.

  1. the first session will be 1 hour to complete an interview about current health and upcoming surgery, a physical assessment, followed by individual exercise demonstration and education.
  2. the second and third session will be follow up sessions to review exercise technique and progress, the presence of abnormal responses, provide encouragement and to address any barriers to activity completion.
  3. the fourth, final session will be at the end of week 3 and will take 30 minutes to review exercise progress, presence of abnormal responses with activity and complete a reassessment of physical function.
* Complete an individualized exercise program 3x/week independently as instructed by the physiotherapist following the initial assessment.
* Complete a home exercise diary to track exercises done and intensity of exercise, in addition to documenting any abnormal responses

For participants who reside in Winnipeg:

* Accelerometers will be delivered to the patients home to wear for:

  1. 7 days prior to the initial assessment
  2. 14 days, from day 8 - 21 of the initial assessment.
* Accelerometer diaries will be provided for participants to complete during the days when the accelerometers are worn.

DETAILED DESCRIPTION:
The study will be a single-centre, prospective, quasi-experimental feasibility study to evaluate a home-based prehab intervention on frail adults undergoing cardiac surgery. The investigators will recruit patients from the St. Boniface Hospital, Winnipeg, Manitoba, an academic, tertiary care hospital.

The goal of this research is to determine the feasibility and safety of a preoperative home-based prehab exercise intervention for frail cardiac surgery patients. The primary research questions include:

1. Will patients display interest in participating in a virtually delivered home-based prehabilitation option compared to in person, center-based recruitment rates?

   a. The investigators hypothesize that patients will display a greater interest in virtually delivered home-based prehabilitation evaluated by recruitment rate being ≥30% (defined as the number of eligible patients that consent to participate).
2. Is the intervention practical, will patients adhere to the prescribed exercises 3 x/week?

   a. The investigators hypothesize that ≥65% of patients will adhere to the exercise protocol.
3. Are the provided exercise images, and live, virtual sessions with the Physiotherapist sufficient to ensure patients are independent with performing the prescribed exercises safely?
4. Are the 4 virtual sessions with the physiotherapist able to be completed in the identified time frames (1 hour for initial assessment and 30 minutes for each of the 3 follow up sessions)?
5. Can the exercise program be completed in the absence of major adverse events?
6. What are the physical activity behaviours of frail patients awaiting cardiac surgery and do they improve with an individualized prehabilitation program?

All patients will participate in a home-based prehab program with individual video sessions via University of Manitoba (UM) Microsoft Teams or UM Zoom, whichever the patient prefers. During a period of three weeks, the patient will meet one on one with a physiotherapist at 4 time points (Figure 1): 1) Initial assessment; 2) within 1 week of the initial assessment; 3) in week two and 4) reassessment of outcomes at the end of three weeks.

The initial session will take an hour and consist of a subjective assessment to confirm the patients scheduled surgery, their past medical history, current medications and inquire about any recent angina or worsening symptoms to determine the patient's medical status to participate. A physical assessment using the Short Physical Performance Battery (SPPB) to stratify patients into an individualized exercise program, followed by exercise demonstration and education. The education will be provided in both verbal and written forms and cover the benefits of exercise on cardiovascular health, the role of balance and strength exercises on improving functional capacity and abnormal responses to exercise with a focus on cardiac symptoms, and an action plan in the event of angina or musculoskeletal discomfort. Patients will be instructed to complete the exercises independently 3x/week in addition to the 4 virtual sessions. The second and third sessions will be 30 minutes in duration and will check in on activity progress, the presence of abnormal responses to exercise, review exercise technique, address barriers and facilitators to activity completion as well as provide support and encouragement for the current level of activity. The final session will take 30 minutes and will review exercise progress and the presence of abnormal responses to exercise followed by a reassessment of physical function. No sessions will be recorded.

The SPPB includes a 3 meter walk test. For patients who do not have a measuring tape to mark the distance within their home, a 3 meter length of yarn will be mailed to them prior to the initial assessment to ensure accuracy.

The 3-week prehabilitation program will focus on balance and strengthening exercises based upon the Otago strength and balance training exercise programme and the Weight-bearing Exercise for Better Balance (WEBB) program. For this study the exercises have been organized into four different levels based on degrees of difficulty, with level 1 being the simplest and level 4 the most challenging. Patients will be stratified into a set of predefined exercises based on the balance component score of the SPPB assessment. Level 1 -SPPB balance score of ≤1; Level 2 - SPPB balance score of 2; Level 3 - SPPB balance score of 3; Level 4 - SPPB balance score of 4. Exercises will be prescribed to be completed three times per week, for three weeks. Patients will be provided with a handout via email discussing the benefits of exercise in cardiovascular health, images with a description of the exercises, signs and symptoms of activity intolerance and an action plan in the event of angina. Additionally, the rating of perceived exertion scale will be provided and explained for patients to best monitor their intensity with the goal of achieving a moderate intensity.

For participants who reside in Winnipeg:

* Accelerometers will be delivered to the patients home to wear for:

  1. 7 days prior to the initial assessment
  2. 14 days, from day 8 - 21 of the initial assessment.
* Accelerometer diaries will be provided for participants to complete during the days when the accelerometers are worn.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥ 18 years of age) undergoing elective isolated coronary artery bypass graft (CABG), aortic valve repair or replacement for moderate aortic stenosis or severe regurgitation, mitral valve repair or replacement for moderate stenosis or severe regurgitation or combined CABG/valve procedures.
2. Patients with a Clinical Frailty Score (CFS) between 3 (managing well) and 6 (living with moderate frailty) as determined by the Cardiac Surgeons or the Nurse Practitioner and/or a score of less than/= 60 on the Short Form 36 Physical Function (SF-36 PF).
3. Patients with an estimated wait time of 3 weeks or longer.
4. Have access to the internet and hardware (smartphone, tablet, computer) to support video telerehabilitation.
5. Have a support person (family member, friend, or caregiver) who is available for all exercise sessions (virtual and independent home exercises). This person should be able to provide technical assistance if needed (help navigate a device to join the telerehabilitation session, set up the device to best view the patient while exercising), is physically capable to stand beside the patient and provide physical assistance if the patient were to lose their balance and is able to respond to any unexpected emergency while the patient is exercising (i.e. provide assistance and/or call 911 if needed).

Exclusion Criteria:

1. Patients who have unstable or recent unstable cardiac syndrome as defined by:

   1. Severe heart failure (NYHA IV) or angina (CCS class IV) symptoms.
   2. Critical left main (LM) coronary disease (>50% stenosis).
   3. Hospitalization for arrhythmias, congestive heart failure (CHF), or acute coronary syndrome (ACS).
2. Patients who have severe left ventricular obstructive disease as defined by:

   a. Severe aortic or mitral stenosis (aortic or mitral valve area <1.0 cm2 or mean gradient > 40 mmHg or > 10 mmHg respectively); or dynamic left ventricular outflow obstruction.
3. Patients who have demonstrated exercise induced ventricular arrhythmias or have experienced a recent hospitalization for arrhythmias.
4. Patients who have cognitive deficits that would preclude prehabilitation.
5. Patients who have physical limitations that would preclude their ability to complete the pre-defined exercises in the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Adverse events related to exercise | Reported at the second virtual visit (in week 1)
  Presence of adverse events related to the exercise intervention
Adverse events related to exercise | Reported at the third virtual visit (in week 2)
  Presence of adverse events related to the exercise intervention
Adverse events related to exercise | Reported at the fourth virtual visit (end of week 3)
  Presence of adverse events related to the exercise intervention
Timing | Reported at initial virtual visit (day 1)
  Length of virtual session
Timing | Reported at second virtual visit (in week 1)
  Length of virtual session
Timing | Reported at third virtual visit (in week 2)
  Length of virtual session
Timing | Reported at final virtual visit (end of week 3)
  Length of virtual session
Exercise technique | Reported at initial virtual session (day 1)
  Number of exercises requiring technique correction
Exercise technique | Reported at second virtual session (in week 1)
  Number of exercises requiring technique correction
Exercise technique | Reported at third virtual session (in week 2)
  Number of exercises requiring technique correction
Exercise technique | Reported at the final virtual session (end of week 3)
  Number of exercises requiring technique correction
Exercise adherence | Reported at second virtual session (in week 1)
  The frequency of home exercises completed and documented in diary
Exercise adherence | Reported at the third virtual session (in week 2)
  The frequency of home exercises completed and documented in diary
Exercise adherence | Reported at the final virtual session (end of week 3)
  The frequency of home exercises completed and documented in diary
Education | Reported at initial virtual session (day 1)
  Frequency of education topics completed
Education | Reported at second virtual session (in week 1)
  Frequency of education topics completed
Education | Reported at the third virtual session (in week 2)
  Frequency of education topics completed
Education | Reported at the final virtual session (end of week 3)
  Frequency of education topics completed
Change in Euro-qol 5 Question-5 Dimension -5 Level (EQ-5D-5L) | Completed at baseline and end of week 3
  The EQ-5D-5L is a quality of life measure that comprises of a short descriptive system questionnaire and a visual analogue scale (EQ-VAS). There are 5 dimensions of health measured to describe current health; 1- Mobility, 2- Self-care, 3 - usual activities, 4 - Pain/discomfort, and 5 - anxiety/depression. Each dimension has 5 descriptive options for each ranging from having no problems/pain (score 1) to being unable to complete activities or being extremely limited by pain or anxiety (score 5). A lower score in each dimension indicates better health.
  The EQ-VAS is a measure of health "today" on a scale of 0 - 100 with 100 being the best health you can imagine and 0 being the worst health you can imagine. A higher score on the EQ-VAS indicates better health.

SECONDARY OUTCOMES:
Change in Short Physical Performance Battery baseline to week 3 | Completed at baseline and end of week 3
  An assessment of lower extremity physical function. It is comprised of three sections, a balance assessment (side by side stance, semi-tandem stance, tandem stance), gait speed, and timed sit to stand. Each of the 3 sections are scored out of 4 points for a maximum score of 12 and a lowest score of 0. The higher the score, the better the physical function.
Change in Duke Activity Status Index baseline to week 3 | Completed at baseline and end of week 3
  The Duke Activity Status Index (DASI) is a functional capacity measure made up of 12 brief questions relating to activities of daily living. The answers correspond to metabolic equivalents required to complete the activities in question. If a patient is unable to complete the activity the score is 0. The lowest score possible is 0, with the maximum score possible being 58.2. The higher the score, the more independent and physically fit the patient is.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Codispodi, BMR PT, Principal Investigator — University of Manitoba; Rakesh Aroroa, MD, Study Director — University of Manitoba; Todd Duhamel, PhD, Study Director — University of Manitoba
Locations (1):
- St Boniface Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to peers for further analysis upon approval by the PI and Co-investigators. Files will be shared by granting access to the de-identified data folders on the University of Manitoba dataverse server. Dataverse is a data repository that contains de-identified data for research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available following publication
Access Criteria: It will be stored on the University of Manitoba's dataverse server

REFERENCES:
- [Background] Steinmetz C, Bjarnason-Wehrens B, Baumgarten H, Walther T, Mengden T, Walther C. Prehabilitation in patients awaiting elective coronary artery bypass graft surgery - effects on functional capacity and quality of life: a randomized controlled trial. Clin Rehabil. 2020 Oct;34(10):1256-1267. doi: 10.1177/0269215520933950. Epub 2020 Jun 16. PMID 32546065
- [Background] Boreskie KF, Hay JL, Kehler DS, Johnston NM, Rose AV, Oldfield CJ, Kumar K, Toleva O, Arora RC, Duhamel TA. Prehabilitation: The Right Medicine for Older Frail Adults Anticipating Transcatheter Aortic Valve Replacement, Coronary Artery Bypass Graft, and Other Cardiovascular Care. Clin Geriatr Med. 2019 Nov;35(4):571-585. doi: 10.1016/j.cger.2019.07.006. Epub 2019 Jul 3. PMID 31543187
- [Background] Yau DKW, Underwood MJ, Joynt GM, Lee A. Effect of preparative rehabilitation on recovery after cardiac surgery: A systematic review. Ann Phys Rehabil Med. 2021 Mar;64(2):101391. doi: 10.1016/j.rehab.2020.03.014. Epub 2020 Oct 14. PMID 32446762
- [Background] Lytwyn J, Stammers AN, Kehler DS, Jung P, Alexander B, Hiebert BM, Dubiel C, Kimber D, Hamm N, Clarke M, Fraser C, Pedreira B, Duhamel TA, Tangri N, Arora RC. The impact of frailty on functional survival in patients 1 year after cardiac surgery. J Thorac Cardiovasc Surg. 2017 Dec;154(6):1990-1999. doi: 10.1016/j.jtcvs.2017.06.040. Epub 2017 Jun 24. PMID 28734627
- [Background] Graham A, Brown CH 4th. Frailty, Aging, and Cardiovascular Surgery. Anesth Analg. 2017 Apr;124(4):1053-1060. doi: 10.1213/ANE.0000000000001560. PMID 27622718
- [Background] Waite I, Deshpande R, Baghai M, Massey T, Wendler O, Greenwood S. Home-based preoperative rehabilitation (prehab) to improve physical function and reduce hospital length of stay for frail patients undergoing coronary artery bypass graft and valve surgery. J Cardiothorac Surg. 2017 Oct 26;12(1):91. doi: 10.1186/s13019-017-0655-8. PMID 29073924
- [Background] Arora RC, Brown CH 4th, Sanjanwala RM, McKelvie R. "NEW" Prehabilitation: A 3-Way Approach to Improve Postoperative Survival and Health-Related Quality of Life in Cardiac Surgery Patients. Can J Cardiol. 2018 Jul;34(7):839-849. doi: 10.1016/j.cjca.2018.03.020. PMID 29960613
- [Background] Engelman DT, Ben Ali W, Williams JB, Perrault LP, Reddy VS, Arora RC, Roselli EE, Khoynezhad A, Gerdisch M, Levy JH, Lobdell K, Fletcher N, Kirsch M, Nelson G, Engelman RM, Gregory AJ, Boyle EM. Guidelines for Perioperative Care in Cardiac Surgery: Enhanced Recovery After Surgery Society Recommendations. JAMA Surg. 2019 Aug 1;154(8):755-766. doi: 10.1001/jamasurg.2019.1153. PMID 31054241
- [Background] Lear SA. The Delivery of Cardiac Rehabilitation Using Communications Technologies: The "Virtual" Cardiac Rehabilitation Program. Can J Cardiol. 2018 Oct;34(10 Suppl 2):S278-S283. doi: 10.1016/j.cjca.2018.07.009. Epub 2018 Jul 18. PMID 30274638
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Arthur HM, Daniels C, McKelvie R, Hirsh J, Rush B. Effect of a preoperative intervention on preoperative and postoperative outcomes in low-risk patients awaiting elective coronary artery bypass graft surgery. A randomized, controlled trial. Ann Intern Med. 2000 Aug 15;133(4):253-62. doi: 10.7326/0003-4819-133-4-200008150-00007. PMID 10929164
- [Background] Sawatzky JA, Kehler DS, Ready AE, Lerner N, Boreskie S, Lamont D, Luchik D, Arora RC, Duhamel TA. Prehabilitation program for elective coronary artery bypass graft surgery patients: a pilot randomized controlled study. Clin Rehabil. 2014 Jul;28(7):648-57. doi: 10.1177/0269215513516475. Epub 2014 Jan 23. PMID 24459173
- [Background] Grant R, Birch N. Otago strength and balance training exercise programme. An information guide for patients. 2021;1-27.
- [Background] Hlatky MA, Boineau RE, Higginbotham MB, Lee KL, Mark DB, Califf RM, Cobb FR, Pryor DB. A brief self-administered questionnaire to determine functional capacity (the Duke Activity Status Index). Am J Cardiol. 1989 Sep 15;64(10):651-4. doi: 10.1016/0002-9149(89)90496-7. PMID 2782256
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Granger CL, Irving L, Antippa P, Edbrooke L, Parry SM, Krishnasamy M, Denehy L. CAPACITY: A physical activity self-management program for patients undergoing surgery for lung cancer, a phase I feasibility study. Lung Cancer. 2018 Oct;124:102-109. doi: 10.1016/j.lungcan.2018.07.034. Epub 2018 Jul 23. PMID 30268446
- [Background] Stammers AN, Kehler DS, Afilalo J, Avery LJ, Bagshaw SM, Grocott HP, Legare JF, Logsetty S, Metge C, Nguyen T, Rockwood K, Sareen J, Sawatzky JA, Tangri N, Giacomantonio N, Hassan A, Duhamel TA, Arora RC. Protocol for the PREHAB study-Pre-operative Rehabilitation for reduction of Hospitalization After coronary Bypass and valvular surgery: a randomised controlled trial. BMJ Open. 2015 Mar 9;5(3):e007250. doi: 10.1136/bmjopen-2014-007250. PMID 25753362